CLINICAL TRIAL: NCT03143816
Title: Study Comparing Prandial Insulin Aspart vs. Technosphere Insulin in Patients With Type 1 Diabetes on Multiple Daily Injections: Investigator-Initiated A Real-life Pilot Study-STAT Study
Acronym: STAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Atlanta Diabetes Associates (Other); University of Southern California (Other); Rainier Clinical Research Center (Other); Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0427
Record Dates: First submitted 2017-05-02; First posted 2017-05-08 (Actual); Results first posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes; time in range; inhaled insulin; continuous glucose monitoring; type 1 diabetes; hypoglycemia; post prandial hypergylcemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Technosphere insulin (TI, Afrezza) -Treatment arm (Active Comparator): Patients who are randomized into the TI arm will be instructed to dose before the meals and take necessary corrections at 1- and 2-hours after meals to optimize PPBG ( post prandial blood glucose)
  Interventions: Drug: Technosphere insulin
- Insulin Aspart ( Novolog) -Control arm (No Intervention): Patients who are randomized into the NL arm will continue using their usual prandial insulin dose before meals.

INTERVENTIONS:
Drug: Technosphere insulin — This multi-center study will enroll 60 patients with T1D, A1c values between 6.5 to 10%. The patients will be randomized in 1:1 fashion to either TI or NL. Patients who are randomized into the NL arm will continue using their usual prandial insulin dose before meals. Patients who are randomized into the TI arm will be instructed to dose before the meals and take necessary corrections at 1- and 2-hours after meals to optimize PPBG (Table 1B). There will be a total of 7 study visits (screening visit, randomization visit, 2 clinic, and 3 phone visits). There will be a 4-week treatment comparison between TI and NL and 1-week of post-study follow up. (Phone visit; Figure-1). Standard lab tests (A1c, complete metabolic panel {CMP}, complete blood count {CBC}) will be performed at the screening visit.
  Arms: Technosphere insulin (TI, Afrezza) -Treatment arm

SUMMARY:
This is an investigator-initiated, prospective, randomized, multicenter, parallel, open-label, pilot clinical trial evaluating the efficacy of TI for PPBG, PPGE, and time-in-range on CGM download in patients with T1D. TI is an inhaled ultra-rapid-acting insulin, approved by the FDA for use in patients with diabetes. This is a pilot, real-life study where patients will continue their routine diabetes care and use post-meal correction dosages as deemed necessary for normalizing PPBG as per the protocol.

This multi-center study will enroll 60 patients with T1D, A1c values between 6.5 to 10%. The patients will be randomized in 1:1 fashion to either TI or NL. Patients who are randomized into the NL arm will continue using their usual prandial insulin dose before meals. Patients who are randomized into the TI arm will be instructed to dose before the meals and take necessary corrections at 1- and 2-hours after meals to optimize PPBG (Table 1B). There will be a total of 7 study visits (screening visit, randomization visit, 2 clinic, and 3 phone visits). There will be a 4-week treatment comparison between TI and NL and 1-week of post-study follow up. (Phone visit; Figure-1). Standard lab tests (A1c, complete metabolic panel {CMP}, complete blood count {CBC}) will be performed at the screening visit.

All patients will use real-time CGM (Dexcom G5®, San Diego, CA), which will be provided at the randomization visit for their day-to-day diabetes care. CGM data will be downloaded at every clinic visit on a secured computer. The data will be analyzed after the study for different primary and secondary end points. All patients will be allowed to keep the CGM after the study is over for their day-to-day diabetes care.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent before any study-related activities,
2. Male or female aged 18-70 years,
3. Type 1 diabetes mellitus (T1D) duration more than six months
4. Treatment with multiple daily injections (MDI) for at least three months before screening visit; stable insulin dose for the last one month,
5. No use of any oral anti-diabetics, any other form of insulin other than mentioned in the protocol, or any other type of injections such as glucagon-like-peptide-1 (GLP-1) analogs, pramlintide or insulin/GLP-1 analog combinations,
6. A1c between 6.5 to 10%,
7. Willingness to routinely collect at least two blood glucose measurements per day needed to calibrate the CGM. Beyond the calibrations, patients may use CGM for necessary action without having to confirm with fingersticks self-monitoring blood glucose (SMBG), as approved by the Food and Drug Administration (FDA),
8. BMI ≤35 kg/m2,
9. Ability and willingness to adhere to the protocol including clinical and phone visits and 4-week-long CGM wear,
10. Using insulin glargine or insulin degludec as basal insulin,
11. Able to use and understand CGM data,
12. Willing to complete phone and clinic visits,
13. Patients who eat three main meals in a day (breakfast, lunch, and dinner),
14. Patients who use insulin-carb ratio for bolus,
15. Ability to speak, read, and write English, and
16. Patients prandial insulin need must be <18 units per meal

Exclusion Criteria:

1. Use of any other diabetic medication other than allowed in the protocol,
2. Pregnant or intention to become pregnant during the study, or not using adequate birth control methods,
3. Severe unexplained hypoglycemia requiring emergency treatment in the previous three months,
4. Use of systemic or inhaled corticosteroids,
5. History of hemoglobinopathies,
6. Diagnosis of anemia,
7. Post-renal transplantation, currently undergoing dialysis, creatinine >2.0 mg/dl or a calculated creatinine clearance of <50 mL/min,
8. Advanced or unstable retinopathy needing laser procedure or vitrectomy,
9. History of pancreatitis,
10. Extensive skin changes/diseases that inhibit wearing a sensor on normal skin,
11. Known allergy to adhesives,
12. Known allergy to study medication,
13. Participation in another investigational study protocol within 30 days before enrollment,
14. Known chronic obstructive pulmonary disease, pulmonary hypertension, asthma, pulmonary fibrosis, or any chronic pulmonary infection, or any systemic disease that primarily affects the lungs. History of any pulmonary nodule will be excluded to participate in the study,
15. Active smokers,
16. Marijuana users,
17. Insulin pump users,
18. Using insulin detemir or NPH as basal insulin, and
19. Any other condition, as determined by the investigator, which could make the subject unsuitable for the trial, impairs the subject's suitability for the trial, or impairs the validity of the informed consent -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Davis Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Publishing the data after the study, presenting at national scientific meetings

REFERENCES:
- [Background] 1. Rathbone M, Hadgraft J, Roberts M, Lane M, Leone-Bay A, Grant M. Technosphere/insulin: mimicking endogenous insulin release. In Modified-Release Drug Delivery Technology. Vol. 2, 2nd ed. Rathbone M, Hadgraft J, Roberts M, Lane M, Eds. New York, Informa Healthcare USA, Inc., 2008, p. 673-679
- [Background] Richardson PC, Boss AH. Technosphere insulin technology. Diabetes Technol Ther. 2007 Jun;9 Suppl 1:S65-72. doi: 10.1089/dia.2007.0212. PMID 17563306
- [Background] https://www.accessdata.fda.gov/drugsatfda_docs/label/2014/022472lbl.pdf, April 2017
- [Background] Bode BW, McGill JB, Lorber DL, Gross JL, Chang PC, Bregman DB; Affinity 1 Study Group. Inhaled Technosphere Insulin Compared With Injected Prandial Insulin in Type 1 Diabetes: A Randomized 24-Week Trial. Diabetes Care. 2015 Dec;38(12):2266-73. doi: 10.2337/dc15-0075. Epub 2015 Jul 15. PMID 26180109
- [Background] Rosenstock J, Lorber DL, Gnudi L, Howard CP, Bilheimer DW, Chang PC, Petrucci RE, Boss AH, Richardson PC. Prandial inhaled insulin plus basal insulin glargine versus twice daily biaspart insulin for type 2 diabetes: a multicentre randomised trial. Lancet. 2010 Jun 26;375(9733):2244-53. doi: 10.1016/S0140-6736(10)60632-0. PMID 20609970
- [Background] Skyler JS, Weinstock RS, Raskin P, Yale JF, Barrett E, Gerich JE, Gerstein HC; Inhaled Insulin Phase III Type 1 Diabetes Study Group. Use of inhaled insulin in a basal/bolus insulin regimen in type 1 diabetic subjects: a 6-month, randomized, comparative trial. Diabetes Care. 2005 Jul;28(7):1630-5. doi: 10.2337/diacare.28.7.1630. PMID 15983312
- [Background] Garg SK, Kelly W, Freson B, Ritchie P. Treat-to-target technosphere insulin study in adult subjects with type 1 diabetes. Poster presented at American Diabetes Association 2011 annual meeting.
- [Derived] Akturk HK, Snell-Bergeon JK, Rewers A, Klaff LJ, Bode BW, Peters AL, Bailey TS, Garg SK. Improved Postprandial Glucose with Inhaled Technosphere Insulin Compared with Insulin Aspart in Patients with Type 1 Diabetes on Multiple Daily Injections: The STAT Study. Diabetes Technol Ther. 2018 Oct;20(10):639-647. doi: 10.1089/dia.2018.0200. Epub 2018 Sep 15. PMID 30207748

RESULTS

PARTICIPANT FLOW:
Groups:
- Technosphere Insulin (TI, Afrezza) -Treatment Arm: There were a total of seven clinic and phone visits during the study period.Patients were randomized 1:1 to TI or insulin aspart group using a blocked design, stratified by screening HbA1c (<8% or >8%).All patients used realtime CGM (continuous glucose monitor) during the study period. Patients randomized to aspart continued the same bolus regimen as used before randomization. If patients were using any other RAIA( rapid acting insulin analog) (other than aspart), they were switched to aspart on the same dose at the randomization visit. Patients in the aspart group were also allowed to change their premeal bolus dose and take postprandial and other correction doses as deemed clinically necessary.
- Aspart ( Control): There were a total of seven clinic and phone visits during the study period.Patients were randomized 1:1 to TI or insulin aspart group using a blocked design, stratified by screening HbA1c (<8% or >8%).All patients used realtime CGM (continuous glucose monitor) during the study period. Patients randomized to aspart continued the same bolus regimen as used before randomization. If patients were using any other RAIA ( rapid acting insulin analog) (other than aspart), they were switched to aspart on the same dose at the randomization visit. Patients in the aspart group were alsoallowed to change their premeal bolus dose and take postprandial and other correction doses as deemed clinically necessary.
Period: Overall Study
Arm/Group | Technosphere Insulin (TI, Afrezza) -Treatment Arm | Aspart ( Control)
Started | 26 | 34
Completed | 22 | 34
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Technosphere Insulin (TI, Afrezza) -Treatment Arm: This group received Technosphere insulin for bolus insulin with meals and corrections
- Insulin Aspart ( Novolog) -Control Arm: This group received insulin aspart for bolus insulin with meals and corrections
- Total: Total of all reporting groups
Arm/Group | Technosphere Insulin (TI, Afrezza) -Treatment Arm | Insulin Aspart ( Novolog) -Control Arm | Total
Number analyzed (Participants) | 26 | 34 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 34 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (16) | 42 (14) | 41 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 16 | 22 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 26 | 34 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 34 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Time in Range (%) (70-180 mg/dl) With TI on CGM
Description: Difference between Time in range for TI group (treatment) and for Aspart group (control)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percent time in range
Groups:
- Insulin Aspart ( Novolog) -Control Arm: Group received insulin aspart as bolus
- Technosphere Insulin (TI, Afrezza) -Treatment Arm: Group received Technosphere insulin as bolus
Arm/Group | Insulin Aspart ( Novolog) -Control Arm | Technosphere Insulin (TI, Afrezza) -Treatment Arm
Number analyzed (Participants) | 34 | 22
percent time in range | 53.5 (1.8) | 58.4 (2.2)

2. Secondary Outcome: Change in Post-prandial Glucose Excursion (mg/dl) (1-4 Hours After Meals) With TI
Description: Difference in postprandial blood glucose between treatment and control group
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Technosphere Insulin (TI, Afrezza) -Treatment Arm: Group using Technosphere insulin
- Insulin Aspart ( Novolog) -Control Arm: Group using novolog ( control ) group
Arm/Group | Technosphere Insulin (TI, Afrezza) -Treatment Arm | Insulin Aspart ( Novolog) -Control Arm
Number analyzed (Participants) | 22 | 34
mg/dl | 45 (6) | 60 (8)

3. Secondary Outcome: Change in Glucose Variability (GV) (mg/dl) (Standard Deviation and/or Coefficient Variation)
Description: Difference of glucose variability metrics between treatment and control groups
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Technosphere Insulin (TI, Afrezza) -Treatment Arm: Group using Technosphere insulin as bolus
- Insulin Aspart ( Novolog) -Control Arm: Group using insulin aspart as bolus
Arm/Group | Technosphere Insulin (TI, Afrezza) -Treatment Arm | Insulin Aspart ( Novolog) -Control Arm
Number analyzed (Participants) | 22 | 34
mg/dl | 57.8 (2.4) | 66.3 (1.9)

4. Secondary Outcome: The Area Under the Curve Calculation (AUC) (Min*mg/dl) in the PPBG and PPGE,
Description: Difference of area under curve between treatment and control groups. ( 0 to 4 hours duration)
Time Frame: 0, 1, 2, 3, 4 hours post-dose at 4 weeks
Measure: Mean (Standard Deviation); unit: min*mg/dl
Groups:
- Technosphere Insulin (TI, Afrezza) -Treatment Arm: The group receiving Technosphere insulin
- Insulin Aspart ( Novolog) -Control Arm: The group receiving insulin aspart (control)
Arm/Group | Technosphere Insulin (TI, Afrezza) -Treatment Arm | Insulin Aspart ( Novolog) -Control Arm
Number analyzed (Participants) | 22 | 34
min*mg/dl | 15020 (560) | 20020 (680)

5. Secondary Outcome: Change in HbA1c (%) in One-month Treatment
Description: Difference in HbA1c between treatment and control group
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percentage (%)
Arm/Group | Technosphere Insulin (TI, Afrezza) -Treatment Arm | Insulin Aspart ( Novolog) -Control Arm
Number analyzed (Participants) | 22 | 34
percentage (%) | 0.25 (0.31) | 0.02 (0.36)

6. Secondary Outcome: Change in Above the Target Time (%) (>180 mg/dl) on CGM
Description: Difference of time above range between treatment and control group
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percent time above target
Arm/Group | Technosphere Insulin (TI, Afrezza) -Treatment Arm | Insulin Aspart ( Novolog) -Control Arm
Number analyzed (Participants) | 22 | 34
percent time above target | 38.1 (0.3) | 41.2 (1.8)

7. Secondary Outcome: Hypoglycemia Frequency (%) (Below the Target <70mg/dl) on CGM
Description: Difference of hypoglycemia frequency between treatment and control groups.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percent time below range
Arm/Group | Technosphere Insulin (TI, Afrezza) -Treatment Arm | Insulin Aspart ( Novolog) -Control Arm
Number analyzed (Participants) | 22 | 34
percent time below range | 2.2 (0.7) | 4.0 (0.6)

ADVERSE EVENTS:
Time Frame: 5 weeks ( 4 weeks treatment and 1 week follow up)
Description: This is a 4-week study, all medications used in this study were FDA approved.
Arm/Group | Technosphere Insulin (TI, Afrezza) -Treatment Arm | Insulin Aspart ( Novolog) -Control Arm
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/34
Other Adverse Events (participants affected / at risk) | 3/26 | 0/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Technosphere Insulin (TI, Afrezza) -Treatment Arm (N=26) | Insulin Aspart ( Novolog) -Control Arm (N=34)
mild cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) — 3 patients reported mild cough in TI group but they continued in the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT03143816/Prot_SAP_001.pdf
  • Informed Consent Form (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT03143816/ICF_002.pdf